CLINICAL TRIAL: NCT01648868
Title: Transcranial Magnetic Stimulation (rTMS) and Autism.Implication of the Superior Temporal Sulcus in Normal and Abnormal Social Perception
Brief Title: Transcranial Magnetic Stimulation (rTMS) and Autism.
Acronym: TMSAUTISME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081232; 2009-A01025-52 (Registry Identifier: ID RCB)
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: TMSAutism; Eye-tracking; Social perception; Social cognition
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Excitatory effects of rTMS (Experimental): Study excitatory effects of rTMS applied to the STS in patients with autism
  Interventions: Device: Transcranial Magnetic Stimulation (rTMS)
- Inhibitory effects of rTMS (Active Comparator): Study inhibitory effects of rTMS applied to the STS in healthy controls
  Interventions: Device: Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (rTMS) — Excitatory effects of Transcranial Magnetic Stimulation (rTMS) applied to the STS in patients with autism.
  Arms: Excitatory effects of rTMS
Device: Transcranial Magnetic Stimulation (rTMS) — Inhibitory effects of Transcranial Magnetic Stimulation (rTMS) applied to the STS in healthy controls
  Arms: Inhibitory effects of rTMS

SUMMARY:
In this protocol we aim to use rTMS to better characterize STS role in normal and abnormal social cognition. With that purpose, we will measure the effect of inhibitory and excitatory rTMS on the fixation time on social scenes (using eye-tracking methodology) or on the ability to recognize human voice/sounds.

DETAILED DESCRIPTION:
Autism is characterized by severe impairments in verbal and non verbal communication and in social interactions. Results from cerebral imaging studies have suggested that abnormalities located on the superior temporal Sulcus (STS) level would be implicated in social impairments in autism. This abnormalities are both anatomical and functional: 1) rest hypoperfusion detected by positron emission tomography (PET); 2) abnormal activation during social tasks (fMRI) and 3) structural abnormalities shown on anatomical MRI. The STS is implicated in social cognition in normal subjects. Our hypothesis is that these anatomo-functional abnormalities would appear very early in brain development and could be one of the first steps in the cascade of neuronal dysfunction in autism. Transcranial Magnetic Stimulation (rTMS) is a technique which is used in cognitive neuroscience research as well as in therapeutic approaches in certain neurological and psychiatry diseases. It consists on applying a magnetic impulse on the brain trough the scalp in a non-invasive and painless by placing a coil on the surface of the head. This magnetic fields induce an electrical field which modifies activity of those neurons inside the magnetic field and induce an electrophysiological change in the target area. This process allows a non-invasive interaction with the human brain in action during focal stimulations. In cognitive neuroscience research, we are interested in the modifications caused by rTMS in cognitive performances in order to better precise the functional role of the target region. The intensity and the frequency of the impulse can be controlled (frequency <1 Hz = inhibitory effect ; frequency > 3 Hz = excitatory effect). The functional characteristics of a given region and it's eventual dysfunctions may be identified thank to the abnormalities in reactivity and cortical connectivity. The goal of this project is to study inhibitory and excitatory effects of rTMS applied to the STS in healthy controls and patients with autism. This effect will be measured by two main parameters of social cognition: 1) visual perception of social scenes, measured by eye-tracking methodology; 2) auditory perception of human voice. We will study 50 healthy voluntaries controls and 50 patients with a non-syndromic autism (18 to 25 years old; IQ > 60), diagnosed by DSM-IV and ADI-R. All participants will undergo an structural MRI and a rTMS session on the STS. In both cases, the STS will be localised based on the structural MRI. The total duration of the rTMS session is about two hours. All data will be analysed by the adapted statistical methods. This study will allow a better understanding of the role of STS in social cognition in healthy subjects as well as it's implication in the social impairments which characterize autism. Finally, the rTMS may become, in a near future, a innovative therapeutic strategy in autism.

ELIGIBILITY:
Inclusion Criteria:

Patients with autism

* Age from 18 to 30 years old
* Autism diagnosed by DSM-IV and ADI-R
* IQ > 60 or able to have an MRI
* Social security registration
* Consent form signed by patient or legal tutor

Healthy controls

* Age from 18 to 30 years old
* Medical exam previous to the interventions
* Social security registration
* Consent form signed

Exclusion Criteria:

All Patients

* Indication against MRI (pace-maker, metallic pieces in the body, working with metals)
* Indications against rTMS (epilepsy, epilepsy family history, craniotomy scarf, pace maker or neuron stimulator, intraocular or intra-cerebral strange metallic piece, cochlear implant, cardiac valve, chirurgical metallic arterial material, metallic material susceptible to concentrate radio-frequency impulse)
* Claustrophobia
* Pregnant woman
* Women in a fertile age with no efficient contraception method
* Use of drugs diminishing cortical excitability
* Participation in another clinical trial that forbids the participation in this one
* Have already being treated by some electrical or magnetic stimulation technique ( transcutaneous or radicular stimulation)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2011-04-06 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Fixation time in eyes, mouth and face areas | 1 day
  Fixation time in eyes, mouth and face areas during the presentation of social scenes

SECONDARY OUTCOMES:
Eye-tracking or voice human perception correlation | 1 day
  Data from eye-tracking or voice human perception (before and after Transcranial Magnetic Stimulation - TMS) will be correlated to different scores of Autism Diagnostic Interview (ADI) : social, communication and repetitive behaviours.
Fractional anisotropy covariation | 1 day
  Covariation of fractional anisotropy (FA) with data from eye-tracking or human voice perception (before and after TMS)
Fractional anisotropy comparison | 1 day
  Comparison of fractional anisotropy (FA) between autistic patients and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie BODDAERT, MD, PhD, Principal Investigator — Necker-Enfants Malades Hospital; Monica ZILBOVICIUS, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saitovitch A, Popa T, Lemaitre H, Rechtman E, Lamy JC, Grevent D, Calmon R, Meunier S, Brunelle F, Samson Y, Boddaert N, Zilbovicius M. Tuning Eye-Gaze Perception by Transitory STS Inhibition. Cereb Cortex. 2016 Jun;26(6):2823-31. doi: 10.1093/cercor/bhw045. Epub 2016 Mar 5. PMID 26946130
- [Background] Saitovitch A, Lemaitre H, Rechtman E, Vincon-Leite A, Calmon R, Grevent D, Dangouloff-Ros V, Brunelle F, Boddaert N, Zilbovicius M. Neural and behavioral signature of human social perception. Sci Rep. 2019 Jun 25;9(1):9252. doi: 10.1038/s41598-019-44977-8. PMID 31239453